CLINICAL TRIAL: NCT00688688
Title: A Randomized, Double-Blind, Parallel Group, Active Controlled, Multi-center Long-term Study to Assess the Safety and Efficacy of the Beta-3 Agonist Mirabegron (YM178) 50 mg qd and 100 mg qd in Subjects With Symptoms of Overactive Bladder
Brief Title: Study to Test the Long Term Safety and Efficacy of the Beta-3 Agonist Mirabegron (YM178) in Patients With Symptoms of Overactive Bladder
Acronym: TAURUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-CL-049; 2007-001452-39 (EudraCT Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Frequency; Overactive Bladder; Urgency; Urinary urge incontinence; Urinary incontinence; Micturition
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence | interventions — mirabegron; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mirabegron 50 mg (Experimental): Participants received mirabegron 50 mg tablets and matching tolterodine extended release (ER) placebo capsules orally once a day for 12 months.
  Interventions: Drug: Mirabegron; Drug: Placebo to Tolterodine
- Mirabegron 100 mg (Experimental): Participants received mirabegron 100 mg tablets and matching tolterodine ER placebo capsules orally once a day for 12 months.
  Interventions: Drug: Mirabegron; Drug: Placebo to Tolterodine
- Tolterodine ER 4 mg (Active Comparator): Participants received tolterodine ER 4 mg capsules and matching mirabegron placebo tablets orally once a day for 12 months.
  Interventions: Drug: Tolterodine; Drug: Placebo to Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Tablets
  Other Names: Myrbetriq; YM178
  Arms: Mirabegron 100 mg; Mirabegron 50 mg
Drug: Tolterodine — Extended release capsules
  Arms: Tolterodine ER 4 mg
Drug: Placebo to Mirabegron — Matching mirabegron placebo tablets.
  Arms: Tolterodine ER 4 mg
Drug: Placebo to Tolterodine — Matching tolterodine placebo capsules.
  Arms: Mirabegron 100 mg; Mirabegron 50 mg

SUMMARY:
The study is intended to test the safety, tolerability, efficacy of two doses of long term once daily (qd) treatment of Mirabegron in patients with symptoms of overactive bladder and secondly to compare these with active comparator.

DETAILED DESCRIPTION:
Patients who completed 178-CL-046 (NCT00689104) or 178-CL-047 (NCT00662909) or new patients could be enrolled in this study if eligible.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to complete the micturition diary and questionnaires correctly
* Patient has symptoms of overactive bladder for ≥ 3 months
* Patient experiences frequency of micturition on average ≥ 8 times per 24-hour period during the 3-day micturition diary period
* Patient must experience at least 3 episodes of urgency (grade 3 or 4) with or without incontinence, during the 3-day micturition diary period

Exclusion Criteria:

* Patient is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential, sexually active and not practicing a highly reliable method of birth control
* Patient has significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor
* Patient has an indwelling catheter or practices intermittent self-catheterization
* Patient has diabetic neuropathy
* Patient has evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Patient receives non-drug treatment including electro-stimulation therapy
* Patient has severe hypertension
* Patient has a known or suspected hypersensitivity to tolterodine, other anticholinergics, YM178, other beta-adrenoreceptor (ß-AR) agonists, or lactose or any of the other inactive ingredients
* Patient has been treated with any investigational drug or device within 30 days (90 days in the UK for all clinical studies except 178-CL-046)
* Patient had an average total daily urine volume > 3000 mL as recorded in the 3-day micturition diary period
* Patient has serum creatinine >150 umol/L, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2x upper limit of normal range (ULN), or gamma-glutamyl transpeptidase (γ-GT) > 3x ULN
* Patient has a clinically significant abnormal electrocardiogram (ECG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2792 (Actual)
Dates: Start 2008-04-25 (Actual); Primary Completion 2010-05-06 (Actual); Study Completion 2010-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (272):
- United States (99):
  - Homewood, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Tucson, Arizona
  - Atherton, California
  - Beverly Hills, California
  - Buena Park, California
  - Fresno, California
  - La Mesa, California
  - Mission Hills, California
  - Newport Beach, California
  - Orange, California
  - Sacramento, California
  - San Bernardino, California
  - San Diego, California
  - Tarzana, California
  - Torrance, California
  - Aurora, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - New Britain, Connecticut
  - Waterbury, Connecticut
  - Aventura, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Wellington, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Coeur d'Alene, Idaho
  - Idaho Falls, Idaho
  - Melrose Park, Illinois
  - Fort Wayne, Indiana
  - Jeffersonville, Indiana
  - Newburgh, Indiana
  - Des Moines, Iowa
  - Wichita, Kansas
  - Greenbelt, Maryland
  - Watertown, Massachusetts
  - North Kansas City, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Endwell, New York
  - Garden City, New York
  - Kingston, New York
  - New York, New York
  - Poughkeepsie, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Wadsworth, Ohio
  - Bethany, Oklahoma
  - Edmond, Oklahoma
  - Bala-Cynwyd, Pennsylvania
  - Jenkintown, Pennsylvania
  - Lancaster, Pennsylvania
  - Reading, Pennsylvania
  - Uniontown, Pennsylvania
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Mountlake Terrace, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
- Woolloongabba, Australia
- Austria (3):
  - Graz
  - Innsbruck
  - Linz
- Minsk, Belarus
- Belgium (8):
  - Antwerp
  - Edegem
  - Ghent
  - Kortrijk
  - Leper
  - Leuven
  - Liège
  - Sint-Truiden
- Canada (21):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - Dartmouth, Nova Scotia
  - Kentville, Nova Scotia
  - Barrie, Ontario
  - Brampton, Ontario
  - Kitchener, Ontario
  - Markham, Ontario
  - Newmarket, Ontario
  - North Bay, Ontario
  - Oshawa, Ontario
  - Saint Denis, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Granby, Quebec
  - Montreal, Quebec
  - Point Claire, Quebec
  - Montreal
- Czechia (8):
  - Brno
  - Mělník
  - Olomouc
  - Ostrava-Poruba
  - Pilsen
  - Prague
  - Štětí
  - Ústí nad Labem
- Denmark (4):
  - Aalborg
  - Aarhus
  - Glostrup Municipality
  - Roskilde
- Finland (4):
  - Helsinki
  - Oulu
  - Tampere
  - Turku
- France (10):
  - Paris, Cedex 10
  - Colmar
  - Marseille
  - Mulhouse
  - Nîmes
  - Orléans
  - Paris-Cedex12
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
- Germany (24):
  - Aichach
  - Bad Ems
  - Bautzen
  - Berlin
  - Duisburg
  - Eisleben Lutherstadt
  - Frankfurt
  - Ganderkesee
  - Hagenow
  - Halle
  - Hamburg
  - Henningsdorf
  - Hettstedt
  - Kiel
  - Koblenz
  - Leipzig
  - Muenchen-Bogenhausen
  - Munich
  - Neustadt in Sachsen
  - Oranienburg
  - Radebeul
  - Sangerhausen
  - Trier
  - Uetersen
- Hungary (7):
  - Budapest
  - Nyíregyháza
  - Sopron
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Tatabánya
- Reykjavik, Iceland
- Ireland (2):
  - Dublin
  - Mullingar
- Italy (10):
  - Bari
  - Catanzaro
  - Genoa
  - Latina
  - Milan
  - Modena
  - Naples
  - Perugia
  - Treviglio
  - Varese
- Latvia (2):
  - Liepāja
  - Riga
- Kaunas, Lithuania
- Netherlands (9):
  - Amsterdam
  - Apeldoorn
  - Eindhoven
  - Enschede
  - Leiden
  - Nijmegen
  - Sneek
  - Tilburg
  - Winterswijk
- Norway (5):
  - Bergen
  - Drammen
  - Hamar
  - Oslo
  - Tønsberg
- Poland (5):
  - Bialystok
  - Lodz
  - Lublin
  - Warsaw
  - Wroclaw
- Portugal (3):
  - Amadora
  - Porto
  - Tomar
- Romania (3):
  - Bucharest
  - Lasi
  - Oradea
- Russia (2):
  - Moscow
  - Saint Petersburg
- Slovakia (5):
  - Martin
  - Poprad
  - Skalica
  - Trenčín
  - Žilina
- South Africa (5):
  - Hatfield
  - Lyttelton
  - Paarl
  - Pietermaritzburg
  - Roodepoort
- Spain (9):
  - Barcelona
  - Bilbao
  - Getafe
  - Madrid
  - Mataró
  - Miranda de Ebro
  - Seville
  - Toledo
  - Valencia
- Sweden (6):
  - Huddinge
  - Örebro
  - Skövde
  - Sonkoping
  - Stockholm
  - Umeå
- Switzerland (2):
  - Frauenfeld
  - Lucerne
- Kiev, Ukraine
- United Kingdom (11):
  - Bristol
  - Chorley
  - Croydon
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Northwood
  - Reading
  - Sheffield
  - Swansea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Background] Chapple CR, Kaplan SA, Mitcheson D, Klecka J, Cummings J, Drogendijk T, Dorrepaal C, Martin N. Randomized double-blind, active-controlled phase 3 study to assess 12-month safety and efficacy of mirabegron, a beta(3)-adrenoceptor agonist, in overactive bladder. Eur Urol. 2013 Feb;63(2):296-305. doi: 10.1016/j.eururo.2012.10.048. Epub 2012 Nov 6. PMID 23195283
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=25

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed the 12-week treatment and safety follow-up periods of studies 178-CL-046 (NCT00689104) or 178-CL-047 (NCT00662909), as well as patients that did not participate in these studies were enrolled into this study if they met all inclusion criteria and none of the exclusion criteria.
Pre-assignment Details: After screening, 2792 patients took placebo run-in study drug in a 2-week, single-blind, placebo run-in period. On completion of the run-in period, 2452 eligible patients were randomly assigned to receive mirabegron 50 mg, or mirabegron 100 mg or tolterodine ER 4 mg once daily for 12 months.
Period: Overall Study
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Started | 815 | 824 | 813
Safety Analysis Set (SAF) | 812 (All randomized patients who took at least 1 dose of double-blind study drug.) | 820 (All randomized patients who took at least 1 dose of double-blind study drug.) | 812 (All randomized patients who took at least 1 dose of double-blind study drug.)
Full Analysis Set (FAS) | 789 (All treated patients with a baseline and at least 1 post-baseline micturition measurement.) | 802 (All treated patients with a baseline and at least 1 post-baseline micturition measurement.) | 791 (All treated patients with a baseline and at least 1 post-baseline micturition measurement.)
Full Analysis Set Incontinence (FAS-I) | 479 (All FAS patients who had at least 1 incontinence episode at Baseline.) | 483 (All FAS patients who had at least 1 incontinence episode at Baseline.) | 488 (All FAS patients who had at least 1 incontinence episode at Baseline.)
Completed | 629 | 645 | 621
Not Completed | 186 | 179 | 192
Not completed — Eligibility criterion not met | 7 | 7 | 10
Not completed — Adverse Event | 52 | 51 | 50
Not completed — Lack of Efficacy | 34 | 25 | 45
Not completed — Withdrawal by Subject | 66 | 75 | 65
Not completed — Lost to Follow-up | 14 | 7 | 7
Not completed — Protocol Violation | 6 | 9 | 11
Not completed — Randomized but never received study drug | 1 | 0 | 0
Not completed — Non-compliance with study procedures | 5 | 3 | 4
Not completed — Taking exclusionary medications | 1 | 0 | 0
Not completed — Site closure | 0 | 1 | 0
Not completed — Violation of exclusion criterion | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg | Total
Number analyzed (Participants) | 812 | 820 | 812 | 2444
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline Measure data are provided for all randomized patients who took at least 1 dose of double-blind study drug (Safety Analysis Set).
  years | 59.2 (12.56) | 60.1 (11.92) | 59.6 (12.47) | 59.6 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 602 | 608 | 600 | 1810
  Male | 210 | 212 | 212 | 634
Type of overactive bladder (OAB) [Number; unit: participants]
  Urge incontinence | 296 | 305 | 317 | 918
  Mixed | 232 | 228 | 210 | 670
  Frequency | 284 | 287 | 285 | 856
Duration of OAB symptoms [Mean (Standard Deviation); unit: months] | 87.4 (96.28) | 87.9 (91.52) | 83.8 (87.34) | 86.4 (91.77)
Summary of previous treatment [Number; unit: participants]
  Placebo | 190 | 174 | 180 | 544
  Mirabegron 50 mg | 170 | 180 | 171 | 521
  Mirabegron 100 mg | 183 | 198 | 197 | 578
  Tolterodine ER 4 mg | 130 | 107 | 108 | 345
  Naive | 139 | 161 | 156 | 456
Mean number of micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions] — The average number of micturitions (urinations) per 24 hours recorded by the patient in a micturition diary for 3 days prior to the Baseline visit.
  micturitions | 11.12 (2.809) | 11.16 (2.917) | 10.94 (2.668) | 11.08 (2.801)
Mean volume voided per micturition [Mean (Standard Deviation); unit: mL] — Recorded by the patient in a micturition diary for 3 days prior to the Baseline visit.
  mL | 160.4 (58.80) | 164.6 (58.62) | 160.8 (56.98) | 162.0 (58.15)
Mean number of urgency episodes (grade 3 or 4) per 24 hours [Mean (Standard Deviation); unit: urgency episodes] — Urgency episodes were those classified by the patient in a 3-day micturition diary as 3 or 4 on the Patient Perception of Intensity of Urgency (PPIUS) scale: 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet.
  urgency episodes | 5.66 (3.601) | 5.61 (3.722) | 5.44 (3.453) | 5.57 (3.594)
Mean level of urgency [Mean (Standard Deviation); unit: scores on a scale] — Average of patients' ratings on the degree of associated urgency for each micturition and/or incontinence episode recorded in a 3-day micturition diary according to the following 5-point categorical scale (Patient Perception of Intensity of Urgency Scale): 0: No urgency; 1: Mild urgency; 2: Moderate urgency, could delay voiding a short while; 3: Severe urgency, could not delay voiding; 4: Urge incontinence, leaked before arriving to the toilet.
  scores on a scale | 2.45 (0.544) | 2.44 (0.525) | 2.43 (0.519) | 2.44 (0.529)
Mean number of nocturia episodes per 24 hours [Mean (Standard Deviation); unit: nocturia episodes] — The average number of times a patient woke at night to urinate (excluding incontinence only episodes) recorded for 3 days prior to the Baseline visit in the patient micturition diary.
  nocturia episodes | 1.83 (1.361) | 1.85 (1.404) | 1.77 (1.388) | 1.82 (1.384)
Mean number of pads used per 24 hours [Mean (Standard Deviation); unit: pads] — Recorded by the patient in a micturition diary for 3 days prior to the Baseline visit.
  pads | 1.06 (1.872) | 0.98 (1.769) | 0.98 (1.759) | 1.01 (1.800)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Severity of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient administered a study drug and which did not necessarily have a causal relationship with the treatment. The investigator assessed the severity of each AE, including abnormal laboratory values, as follows:
  Mild: No disruption of normal daily activities; Moderate: Affected normal daily activities; Severe: Inability to perform daily activities.
Time Frame: From the first dose of double-blind study drug up until 30 days after the last dose of study drug, up to 13 months.
Population: The number of participants analyzed represents the Safety Analysis Set (SAF), including all randomized patients who took at least one dose of double-blind study drug.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 812 | 820 | 812
participants
  Mild adverse events | 222 | 240 | 251
  Moderate adverse events | 212 | 211 | 218
  Severe adverse events | 51 | 52 | 39

2. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was derived from the number of times a patient urinates (excluding incontinence only episodes) per day recorded by the patient in a micturition diary for 3-days prior to clinic visits at Baseline and months 1, 3, 6, 9 and 12/end of treatment. Least squares (LS) means were generated from the analysis of covariance (ANCOVA) model with treatment group, previous study history, gender and geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all randomized patients who took at least 1 dose of double-blind study drug with a baseline and at least 1 post baseline micturition measurement in the visit diary. N is the number of patients included in the analysis at each time point. Last observation carried forward (LOCF) was used for the Final Visit analysis.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
micturitions
  Month 1 [N=786; 797; 786] | -0.94 (0.069) | -1.10 (0.068) | -1.02 (0.069)
  Month 3 [N=742; 741; 735] | -1.13 (0.079) | -1.46 (0.079) | -1.27 (0.080)
  Month 6 [N=684; 705; 684] | -1.25 (0.083) | -1.43 (0.082) | -1.30 (0.083)
  Month 9 [N=656; 667; 645] | -1.33 (0.086) | -1.37 (0.086) | -1.38 (0.087)
  Month 12 [N=627; 642; 623] | -1.30 (0.089) | -1.46 (0.088) | -1.50 (0.089)
  Final Visit (LOCF) [N=789; 802; 791] | -1.27 (0.083) | -1.41 (0.082) | -1.39 (0.083)

3. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per day was derived from the number of incontinence episodes recorded by the patient in a micturition diary for 3-days prior to clinic visits at Baseline and months 1, 3, 6, 9 and 12/end of treatment. Least squares (LS) means were generated from the analysis of covariance (ANCOVA) model with treatment group, previous study history, gender and geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set-Incontinence included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary & who had at least 1 incontinence episode at baseline. N is the number of patients included at each time point. LOCF was used for the Final Visit analysis.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 479 | 483 | 488
incontinence episodes
  Month 1 [N=478; 479; 485] | -0.94 (0.079) | -1.03 (0.079) | -0.96 (0.078)
  Month 3 [N=447; 443; 452] | -1.10 (0.083) | -1.28 (0.084) | -1.09 (0.083)
  Month 6 [N=409; 428; 418] | -1.11 (0.088) | -1.27 (0.086) | -1.17 (0.087)
  Month 9 [N=387; 402; 391] | -1.17 (0.083) | -1.32 (0.082) | -1.26 (0.083)
  Month 12 [N=370; 387; 379] | -1.14 (0.094) | -1.19 (0.092) | -1.36 (0.093)
  Final Visit (LOCF) [N=479; 483; 488] | -1.01 (0.087) | -1.24 (0.086) | -1.26 (0.086)

4. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Volume Voided Per Micturition
Description: The average volume voided per micturition was calculated from the volume of each micturition measured by the patient and recorded in a micturition diary for 3 days prior to clinic visits at Baseline and months 1, 3, 6, 9 and 12/end of treatment. LS means were generated from the ANCOVA model with treatment group, previous study history, gender and geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
mL
  Month 1 [N=785; 797; 786] | 12.1 (1.31) | 16.7 (1.30) | 16.0 (1.31)
  Month 3 [N=741; 741; 735] | 14.8 (1.50) | 20.4 (1.50) | 17.4 (1.51)
  Month 6 [N=684; 705; 684] | 18.6 (1.69) | 23.0 (1.66) | 18.8 (1.69)
  Month 9 [N=655; 667; 645] | 20.5 (1.78) | 23.5 (1.77) | 17.9 (1.80)
  Month 12 [N=626; 642; 623] | 18.5 (1.86) | 24.3 (1.83) | 18.9 (1.86)
  Final Visit (LOCF) [N=789; 802; 791] | 17.5 (1.65) | 21.5 (1.63) | 18.1 (1.64)

5. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: The involuntary leakage of urine accompanied or immediately proceeded by urgency, derived from the number of incontinence episodes classified by the patient in a 3-day micturition diary as 3 or 4 on the Patient Perception of Intensity of Urgency Scale: 0=No urgency; 1=Mild urgency; 2=Moderate urgency, could postpone voiding a short time; 3=Severe urgency, could not postpone voiding; 4=Urge incontinence, leaked before arriving to toilet. LS means are from the ANCOVA model with treatment group, previous study history, gender and geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set-Incontinence included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary & who had at least 1 urgency incontinence episode at baseline. N is the number of patients included at each time point. LOCF is used for the Final Visit.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 479 | 483 | 488
urgency incontinence episodes
  Month 1 [N=471; 467; 471] | -0.92 (0.072) | -1.04 (0.073) | -0.95 (0.072)
  Month 3 [N=441; 432; 440] | -1.05 (0.077) | -1.23 (0.078) | -1.06 (0.077)
  Month 6 [N=404; 417; 408] | -1.13 (0.080) | -1.32 (0.079) | -1.11 (0.080)
  Month 9 [N=382; 392; 382] | -1.13 (0.077) | -1.33 (0.076) | -1.25 (0.077)
  Month 12 [N=366; 377; 371] | -1.17 (0.087) | -1.20 (0.085) | -1.29 (0.086)
  Final Visit (LOCF) [N=472; 471; 474] | -1.01 (0.082) | -1.23 (0.082) | -1.21 (0.081)

6. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Number of Urgency Episodes (Grade 3 and/or 4) Per 24 Hours
Description: The average number of urgency episodes (the sudden, compelling desire to pass urine that is difficult to defer) derived from episodes classified by the patient in a 3-day micturition diary as 3 or 4 on the Patient Perception of Intensity of Urgency Scale: 0=No urgency; 1=Mild urgency; 2=Moderate urgency, could delay voiding a short time; 3=Severe urgency, could not delay voiding; 4=Urge incontinence, leaked before arriving to the toilet. LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary. This analysis includes patients with at least 1 urgency episode at Baseline. N is the number of patients included at each time point. LOCF is used for the Final Visit.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
urgency episodes
  Month 1 [N=783; 791; 780] | -1.30 (0.092) | -1.31 (0.091) | -1.11 (0.092)
  Month 3 [N=738; 737; 733] | -1.37 (0.103) | -1.83 (0.103) | -1.55 (0.103)
  Month 6 [N=683; 701; 680] | -1.75 (0.108) | -1.95 (0.106) | -1.63 (0.108)
  Month 9 [N=653; 665; 643] | -1.77 (0.114) | -1.71 (0.113) | -1.78 (0.115)
  Month 12 [N=621; 637; 621] | -1.81 (0.116) | -1.79 (0.115) | -1.89 (0.116)
  Final Visit (LOCF) [N=788; 799; 788] | -1.62 (0.108) | -1.80 (0.107) | -1.63 (0.108)

7. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Level of Urgency
Description: Average of patients' ratings on the degree of urgency associated with each micturition and/or incontinence episode recorded in a 3-day micturition diary according to the Patient Perception of Intensity of Urgency Scale: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could delay voiding a short while; 3 = Severe urgency, could not delay voiding; 4 = Urge incontinence, leaked before arriving to the toilet. LS means are generated from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug with a baseline and at least 1 postbaseline micturition measurement in the visit diary. N is the number of patients included at each time point. LOCF is used for the Final Visit analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
scores on a scale
  Month 1 [N=784; 793; 780] | -0.18 (0.016) | -0.19 (0.016) | -0.17 (0.016)
  Month 3 [N=739; 738; 733] | -0.21 (0.019) | -0.28 (0.019) | -0.24 (0.019)
  Month 6 [N=684; 702; 680] | -0.29 (0.021) | -0.32 (0.021) | -0.27 (0.021)
  Month 9 [N=654; 666; 643] | -0.30 (0.022) | -0.30 (0.022) | -0.31 (0.022)
  Month 12 [N=622; 638; 621] | -0.33 (0.023) | -0.31 (0.023) | -0.32 (0.023)
  Final Visit (LOCF) [N=789; 801; 788] | -0.29 (0.020) | -0.29 (0.020) | -0.27 (0.020)

8. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in the Mean Number of Pads Used Per 24 Hours
Description: The average number of times a patient records a new pad used per day during the 3-day micturition diary period.
  LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary. This analysis includes patients who had at least 1 use of a pad at Baseline. N is the number of patients included at each time point. LOCF is used for the Final Visit
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
pads
  Month 1 [N=324; 305; 313] | -0.75 (0.084) | -0.79 (0.086) | -0.79 (0.085)
  Month 3 [N=307; 280; 286] | -0.80 (0.093) | -0.94 (0.097) | -0.95 (0.096)
  Month 6 [N=277; 271; 264] | -0.88 (0.097) | -0.94 (0.098) | -0.99 (0.099)
  Month 9 [N=264; 255; 250] | -0.99 (0.092) | -0.96 (0.094) | -0.99 (0.094)
  Month 12 [N=254; 247; 241] | -0.87 (0.100) | -0.92 (0.101) | -1.13 (0.102)
  Final Visit (LOCF) [N=325; 307; 314] | -0.81 (0.089) | -0.88 (0.092) | -1.02 (0.090)

9. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Mean Number of Nocturia Episodes Per 24 Hours
Description: Nocturia is defined as waking at night one or more times to void. The average number of times a patient urinated (excluding incontinence only episodes) during sleeping time per day was derived from the 3-day patient micturition diary.
  LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary. This analysis includes patients with at least 1 nocturia episode at Baseline. N is the number of patients included at each time point. LOCF is used for the Final Visit.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
nocturia episodes
  Month 1 [N=690; 698; 690] | -0.26 (0.034) | -0.29 (0.033) | -0.29 (0.034)
  Month 3 [N=654; 651; 643] | -0.41 (0.037) | -0.45 (0.037) | -0.37 (0.037)
  Month 6 [N=604; 618; 602] | -0.42 (0.041) | -0.38 (0.040) | -0.35 (0.041)
  Month 9 [N=580; 583; 567] | -0.50 (0.040) | -0.41 (0.040) | -0.39 (0.040)
  Month 12 [N=554; 562; 550] | -0.48 (0.042) | -0.40 (0.041) | -0.46 (0.042)
  Final Visit (LOCF) [N=693; 703; 693] | -0.46 (0.038) | -0.39 (0.038) | -0.43 (0.038)

10. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes at Months 1, 3, 6, 9 and 12 and the Final Visit
Description: The percentage of participants with no incontinence episodes for the 3 days prior to each clinic visit derived from the micturition diary recorded by the patient.
Time Frame: Months 1, 3, 6, 9 and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 479 | 483 | 488
percentage of participants
  Month 1 [N=478; 479; 485] | 35.4 | 36.7 | 33.4
  Month 3 [N=447; 443; 452] | 40.9 | 45.4 | 39.2
  Month 6 [N=409; 428; 418] | 43.3 | 45.1 | 43.5
  Month 9 [N=387; 402; 391] | 47.5 | 46.8 | 44.2
  Month 12 [N=370; 387; 379] | 47.8 | 47.5 | 49.1
  Final Visit (LOCF) [N=479; 483; 488] | 43.4 | 45.8 | 45.1

11. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction in Incontinence Episodes at Months 1, 3, 6, 9 and 12 and the Final Visit
Description: The percentage of participants with at least a 50% decrease from baseline in mean number of incontinence episodes per 24 hours during the 3 days prior to each clinic visit derived from the patient micturition diary.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 479 | 483 | 488
percentage of participants
  Month 1 [N=478; 479; 485] | 58.2 | 57.0 | 56.3
  Month 3 [N=447; 443; 452] | 61.7 | 66.1 | 61.5
  Month 6 [N=409; 428; 418] | 65.5 | 66.8 | 63.9
  Month 9 [N=387; 402; 391] | 65.6 | 67.2 | 66.0
  Month 12 [N=370; 387; 379] | 67.6 | 68.5 | 71.2
  Final Visit (LOCF) [N=479; 483; 488] | 63.7 | 66.3 | 66.8

12. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Symptom Bother Score
Description: Overactive bladder symptoms were assessed using the symptom bother scale of the overactive bladder questionnaire. The symptom bother scale consists of 8 questions answered by the patient on a scale from 1-6. The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. A negative change from Baseline in symptom bother score indicates improvements.
  LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary. N is the number of patients included at each time point. LOCF is used for the Final Visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
scores on a scale
  Month 1 [N=775; 784; 771] | -10.5 (0.55) | -12.5 (0.55) | -11.5 (0.55)
  Month 3 [N=736; 733; 739] | -13.4 (0.61) | -16.1 (0.61) | -13.5 (0.60)
  Month 6 [N=680; 699; 682] | -14.5 (0.65) | -16.5 (0.64) | -14.6 (0.64)
  Month 9 [N=649; 661; 639] | -14.2 (0.68) | -15.6 (0.68) | -14.3 (0.69)
  Month 12 [N=622; 636; 612] | -14.1 (0.70) | -15.7 (0.69) | -16.3 (0.71)
  Final Visit (LOCF) [N=779; 795; 781] | -13.1 (0.65) | -14.8 (0.65) | -14.3 (0.65)

13. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in Health-related Quality of Life (HRQL) Total Score
Description: Health-related quality of life was assessed by the HRQL subscales (coping, concern, sleep and social interaction) of the overactive bladder questionnaire (OABq). The HRQL total score was calculated by adding the 4 HRQL subscale scores, and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from Baseline in HRQL score indicates improvements.
  LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
scores on a scale
  Month 1 [N=774; 787; 773] | 7.7 (0.48) | 8.9 (0.48) | 8.9 (0.48)
  Month 3 [N=736; 740; 739] | 9.9 (0.54) | 11.9 (0.54) | 10.6 (0.54)
  Month 6 [N=681; 700; 686] | 11.7 (0.56) | 12.9 (0.56) | 11.6 (0.56)
  Month 9 [N=650; 667; 644] | 11.3 (0.60) | 12.2 (0.59) | 12.4 (0.60)
  Month 12 [N=619; 640; 613] | 11.7 (0.62) | 12.6 (0.61) | 13.2 (0.62)
  Final Visit (LOCF) [N=779; 798; 783] | 10.7 (0.58) | 11.7 (0.57) | 11.4 (0.58)

14. Secondary Outcome: Change From Baseline to Month 12 and Final Visit in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. A negative change from Baseline score indicates improvement.
  LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Month 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug with a baseline & at least 1 postbaseline micturition measurement in the visit diary. The number of participants included at each time point (N) only includes those with baseline and post-baseline values. LOCF is used for the Final Visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
scores on a scale
  Month 12 [N=601; 616; 611] | -0.8 (0.04) | -0.9 (0.04) | -0.9 (0.04)
  Final Visit (LOCF) [N=655; 673; 673] | -0.8 (0.04) | -0.9 (0.04) | -0.8 (0.04)

15. Secondary Outcome: Change From Baseline to Month 12 and Final Visit in Treatment Satisfaction-visual Analog Scale (TS-VAS)
Description: The TS-VAS is a visual analog scale (VAS) that asks patients to rate their satisfaction with treatment by placing a vertical mark on a 10 cm line where the endpoints are labeled 'No, not at all' on the left (=0) to 'Yes, completely satisfied' on the right (=10). A positive change from baseline indicates improvement. LS means are from an ANCOVA model with treatment group, previous study history, gender & geographical regions as fixed factors and baseline as a covariate.
Time Frame: Baseline and Month 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
scores on a scale
  Month 12 [N=599; 620; 613] | 2.27 (0.175) | 2.27 (0.172) | 2.52 (0.173)
  Final Visit (LOCF) [N=654; 676; 676] | 2.08 (0.167) | 2.11 (0.164) | 2.27 (0.164)

16. Secondary Outcome: Change From Baseline to Months 3, 6, 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with work productivity in the last 7 days. Percent of work time missed is derived from the number of hours of work missed due to OAB symptoms as a percentage of total hours that should have been worked. A higher percentage indicates more hours missed. A negative change from baseline indicates improvement.
Time Frame: Baseline and Months 3, 6 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary. The number of patients at each time point (N) includes those with both baseline and post-baseline values who were employed. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: Percent work time missed
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
Percent work time missed
  Month 3 [N=215; 217; 211] | -0.06 (7.48) | -1.0 (9.41) | -0.6 (12.38)
  Month 6 [N=183; 203; 200] | -1.3 (6.80) | -1.5 (10.62) | -0.7 (6.26)
  Month 12 [N=181; 185; 188] | -0.5 (9.55) | -0.8 (12.39) | -1.2 (8.08)
  Final Visit (LOCF) [N=245; 256; 249] | -0.5 (8.98) | -0.9 (10.98) | -0.8 (11.37)

17. Secondary Outcome: Change From Baseline to Months 3, 6, 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Impairment While Working
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with work productivity in the last 7 days. Percent impairment while working was derived from the patient's assessment of the degree to which OAB affected their productivity while working. A higher percentage indicates greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent impairment while working
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
Percent impairment while working
  Month 3 [N=233; 236; 231] | -10.6 (23.36) | -9.9 (23.65) | -10.9 (22.56)
  Month 6 [N=207; 216; 213] | -13.0 (22.44) | -11.9 (21.88) | -11.1 (22.21)
  Month 12 [N=194; 196; 201] | -11.9 (24.37) | -14.4 (26.00) | -12.3 (24.60)
  Final Visit (LOCF) [N=261; 272; 265] | -10.9 (24.51) | -11.8 (25.12) | -10.6 (24.34)

18. Secondary Outcome: Change From Baseline to Months 3, 6, 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Overall Work Impairment
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with work productivity in the last 7 days. Percent overall work impairment takes into account both hours missed due to OAB symptoms and the patient's assessment of the degree to which OAB affected their productivity while working. A higher percentage indicates greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent overall work impairment
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
Percent overall work impairment
  Month 3 [N=208; 208; 204] | -11.4 (23.92) | -10.9 (24.50) | -11.0 (23.10)
  Month 6 [N=181; 195; 193] | -12.4 (22.29) | -13.0 (23.99) | -11.1 (22.48)
  Month 12 [N=175; 177; 183] | -11.5 (25.36) | -14.1 (27.02) | -13.6 (25.75)
  Final Visit (LOCF) [N=240; 250; 244] | -11.2 (25.21) | -12.4 (25.56) | -11.5 (24.74)

19. Secondary Outcome: Change From Baseline to Months 3, 6, 12 and Final Visit in Work Productivity and Activity Impairment (WPAI): Percent Activity Impairment
Description: The Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) questionnaire was used to assess the degree and extent to which overactive bladder (OAB) symptoms interfered with daily activities over the last 7 days. Percent activity impairment is derived from the patient's assessment of the degree to which OAB affected their regular daily activities. A higher percentage indicates greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline and Months 3, 6 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary. The number of patients at each time point (N) includes those with both baseline and post-baseline value. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
Percent activity impairment
  Month 3 [N=691; 690; 692] | -12.0 (24.21) | -13.7 (25.75) | -12.3 (25.34)
  Month 6 [N=640; 663; 651] | -14.0 (25.47) | -15.6 (26.38) | -13.4 (26.25)
  Month 12 [N=582; 603; 598] | -13.3 (26.50) | -15.2 (28.84) | -15.0 (28.07)
  Final Visit (LOCF) [N=728; 737; 733] | -12.5 (26.37) | -13.9 (28.53) | -12.8 (28.10)

20. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Mobility Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and evaluating health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no problems in walking about; I have some problems in walking about; I am confined to bed.
  In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Month 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug and had a baseline and at least 1 postbaseline micturition measurement in the visit diary. LOCF was used for this analysis.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
participants
  No problem -> No problem | 567 | 601 | 573
  No problem -> Some problems | 36 | 42 | 39
  No problem -> Confined to bed | 1 | 1 | 0
  No problem -> Missing data | 4 | 3 | 2
  Some problems -> No problems | 64 | 55 | 62
  Some problems -> Some problems | 105 | 97 | 106
  Some problems -> Confined to bed | 1 | 0 | 0
  Some problems -> Missing data | 0 | 1 | 2
  Confined to bed -> No problems | 0 | 1 | 0
  Confined to bed -> Some problems | 0 | 0 | 0
  Confined to bed -> Confined to bed | 0 | 0 | 0
  Confined to bed -> Missing data | 0 | 0 | 0
  Missing data -> No problem | 11 | 1 | 7
  Missing data -> Some problems | 0 | 0 | 0
  Missing data -> Confined to bed | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Self-Care Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and evaluating health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no problems with self-care; I have some problems washing or dressing myself; I am unable to wash or dress myself. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Month 12
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
participants
  No problem -> No problem | 718 | 735 | 720
  No problem -> Some problems | 16 | 15 | 23
  No problem -> Unable to wash or dress myself | 1 | 0 | 3
  No problem -> Missing data | 4 | 4 | 4
  Some problems -> No problems | 19 | 19 | 13
  Some problems -> Some problems | 18 | 25 | 20
  Some problems -> Unable to wash or dress myself | 0 | 0 | 0
  Some problems -> Missing data | 0 | 0 | 0
  Unable to wash or dress myself -> No problems | 0 | 2 | 0
  Unable to wash or dress myself -> Some problems | 0 | 1 | 0
  Unable to wash or dress -> Unable to wash or dress | 0 | 0 | 0
  Unable to wash or dress myself -> Missing data | 0 | 0 | 0
  Missing data -> No problem | 13 | 1 | 8
  Missing data -> Some problems | 0 | 0 | 0
  Missing data -> Unable to wash or dress myself | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Usual Activities Score
Description: The EQ-5D is a standardized, nondisease-specific instrument for describing health status. Participants were asked which statement best describes their health state with regard to usual activities (work, study or leisure): I have no problems performing my usual activities; I have some problems performing my usual activities; I am unable to perform my usual activities. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available at that Visit.
Time Frame: Baseline and Month 12
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
participants
  No problem -> No problem | 536 | 569 | 542
  No problem -> Some problems | 40 | 55 | 53
  No problem -> Unable to perform usual activities | 2 | 1 | 2
  No problem -> Missing data | 3 | 1 | 1
  Some problems -> No problems | 97 | 88 | 96
  Some problems -> Some problems | 94 | 76 | 79
  Some problems-> Unable to perform usual activities | 1 | 2 | 1
  Some problems -> Missing data | 1 | 2 | 3
  Unable to perform usual activities -> No problems | 0 | 2 | 0
  Unable to perform usual activities-> Some problems | 2 | 4 | 5
  Unable to perform -> Unable to perform | 2 | 0 | 1
  Unable to perform usual activities -> Missing data | 10 | 2 | 7
  Missing data -> No problem | 1 | 0 | 1
  Missing data -> Some problems | 0 | 0 | 0
  Missing data -> Unable to perform usual activities | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Pain/Discomfort Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and evaluating health status. Participants were asked to indicate which of the following statements best describes their health state:
  I have no pain or discomfort; I have moderate pain or discomfort; I have extreme pain or discomfort. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Month 12
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
participants
  No pain -> No pain | 398 | 396 | 398
  No pain -> Moderate pain | 54 | 69 | 63
  No pain -> Extreme pain | 4 | 2 | 4
  No pain -> Missing data | 4 | 2 | 2
  Moderate pain -> No pain | 104 | 107 | 105
  Moderate pain -> Moderate pain | 173 | 196 | 182
  Moderate pain -> Extreme pain | 14 | 5 | 8
  Moderate pain -> Missing data | 1 | 2 | 2
  Extreme pain -> No pain | 3 | 4 | 4
  Extreme pain -> Moderate pain | 13 | 6 | 9
  Extreme pain -> Extreme pain | 10 | 10 | 8
  Extreme pain -> Missing data | 0 | 0 | 0
  Missing data-> No pain | 8 | 3 | 6
  Missing data -> Moderate pain | 3 | 0 | 0
  Missing data -> Extreme pain | 0 | 0 | 0
  Missing data -> Missing data | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline to Final Visit in European Quality of Life-5 Dimensions (EQ-5D) Anxiety/Depression Score
Description: The EQ-5D is an international, standardized, nondisease-specific (i.e., generic) instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state:
  I am not anxious or depressed; I am moderately anxious or depressed; I am extremely anxious or depressed. In the table below, each row title lists Baseline health status first followed by Final Visit health status and reports the number of patients in that category. Missing data indicates patients with no data available for that Visit.
Time Frame: Baseline and Month 12
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
participants
  Not anxious -> Not anxious | 413 | 453 | 429
  Not anxious -> Moderately anxious | 43 | 34 | 43
  Not anxious -> Extremely anxious | 3 | 3 | 1
  Not anxious -> Missing data | 3 | 1 | 2
  Moderately anxious -> Not anxious | 108 | 99 | 105
  Moderately anxious -> Moderately anxious | 174 | 181 | 169
  Moderately anxious -> Extremely anxious | 7 | 9 | 11
  Moderately anxious -> Missing data | 1 | 2 | 2
  Extremely anxious -> Not anxious | 3 | 5 | 3
  Extremely anxious -> Moderately anxious | 8 | 9 | 14
  Extremely anxious -> Extremely anxious | 15 | 5 | 6
  Extremely anxious -> Missing data | 0 | 0 | 0
  Missing data -> Not anxious | 7 | 0 | 3
  Missing data -> Moderately anxious | 4 | 1 | 2
  Missing data -> Extremely anxious | 0 | 0 | 1
  Missing data -> Missing data | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline to Months 1, 3, 6, 9, 12 and Final Visit in the European Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D is an international, standardized, generic instrument for describing and evaluating health status. Health status is assessed by patients evaluating their health on a vertical, visual analog scale from 0 to 100 where the endpoints are labeled 'Worst imaginable health state' (=0) and 'Best imaginable health state' (=100). On the EQ-5D VAS, a positive change from Baseline indicates improvement.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12
Population: The full analysis set included all patients who took at least 1 dose of double-blind study drug & had a baseline & at least 1 postbaseline micturition measurement in the visit diary. The number of patients at each time point (N) includes those with both baseline and post-baseline values. LOCF was used for the Final Visit analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
scores on a scale
  Month 1 [N=767; 787; 770] | 3.8 (12.85) | 3.9 (13.64) | 3.1 (12.78)
  Month 3 [N=734; 740; 731] | 5.0 (15.33) | 5.4 (15.27) | 4.3 (13.48)
  Month 6 [N=676; 697; 678] | 6.5 (16.97) | 6.4 (16.54) | 5.2 (15.40)
  Month 9 [N=645; 665; 637] | 6.6 (17.52) | 6.5 (16.55) | 6.3 (15.91)
  Month 12 [N=615; 637; 612] | 8.2 (17.39) | 6.8 (17.56) | 7.9 (16.48)
  Final Visit (LOCF) [N=776; 797; 777] | 6.8 (17.47) | 5.9 (17.35) | 6.0 (16.64)

26. Secondary Outcome: Change From Baseline to Months 3, 6, 12 and Final Visit in Number of Non-study Related Visits to Physician
Description: The number of times the patient visited a physician's office during the 4 weeks prior to each study visit (excluding study visits) because of the patient's bladder condition.
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Physician visits
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
Physician visits
  Month 3 [N=748; 750; 744] | 0.0 (0.22) | 0.0 (0.15) | 0.0 (0.14)
  Month 6 [N=690; 705; 687] | 0.0 (0.17) | 0.0 (0.13) | 0.0 (0.18)
  Month 12 [N=628; 640; 622] | 0.0 (0.25) | 0.0 (0.13) | 0.0 (0.11)
  Final Visit (LOCF) [N=773; 769; 760] | 0.0 (0.25) | 0.0 (0.15) | 0.0 (0.14)

27. Secondary Outcome: Percentage of Participants With Improvement in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. Improvement was defined as at least a one point improvement from Baseline to post-baseline and a major improvement was defined as at least a two point improvement from Baseline to post-baseline in PPBC score.
Time Frame: Baseline and Month 12
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 789 | 802 | 791
percentage of participants
  Improvement: Month12 [N=616; 630; 620] | 55.7 | 60.6 | 56.6
  Improvement: Final Visit [N=671; 688; 684] | 52.9 | 59.6 | 54.4
  Major Improvement: Month 12 [N=616; 630; 620] | 27.4 | 29.7 | 28.2
  Major Improvement: Final Visit [N=671; 688; 684] | 26.2 | 28.2 | 26.6

28. Secondary Outcome: Safety as Assessed by Adverse Events (AEs), Vital Signs, Laboratory Tests, Physical Examination and Electrocardiogram
Description: An abnormality identified during a medical test was defined as an AE if the abnormality induced clinical signs or symptoms, required active intervention, interruption or discontinuation of study drug or was clinically significant. The Investigator assessed each AE for causal relationship (not related, possible or probable) to study drug. A serious AE (SAE) was any untoward medical occurrence that: resulted in death, was life-threatening, resulted in significant disability/incapacity or congenital anomaly/birth defect, required or prolonged hospitalization or was a medically important event.
  The data reported represent the number of participants with adverse events in each category.
Time Frame: From the first dose of double-blind study drug up until 30 days after the last dose of study drug, up to 13 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 812 | 820 | 812
participants
  Adverse events | 485 | 503 | 508
  Treatment-related adverse events (TRAEs) | 213 | 192 | 224
  Deaths | 2 | 0 | 2
  Serious adverse events (SAEs) | 42 | 51 | 44
  Treatment-related serious adverse events | 10 | 4 | 5
  AEs leading to study drug discontinuation | 48 | 50 | 46
  TRAEs leading to study drug discontinuation | 35 | 29 | 31

ADVERSE EVENTS:
Time Frame: Adverse events starting or worsening in the period from first double-blind study drug intake until 30 days after last double-blind study drug intake.
Arm/Group | Mirabegron 50 mg | Mirabegron 100 mg | Tolterodine ER 4 mg
Serious Adverse Events (participants affected / at risk) | 42/812 | 51/820 | 44/812
Other Adverse Events (participants affected / at risk) | 136/812 | 137/820 | 181/812
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 50 mg (N=812) | Mirabegron 100 mg (N=820) | Tolterodine ER 4 mg (N=812)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0
Cystocele repair (Surgical and medical procedures) | 0 | 1 | 0
Gastrectomy (Surgical and medical procedures) | 1 | 0 | 0
Gastric bypass (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 0
Uterine prolapse repair (Surgical and medical procedures) | 0 | 1 | 0
Cystopexy (Surgical and medical procedures) | 0 | 0 | 1
Foot operation (Surgical and medical procedures) | 0 | 0 | 1
Spinal laminectomy (Surgical and medical procedures) | 0 | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Intestinal gangrene (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral circulatory failure (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Global amnesia (Nervous system disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Ischaemia (Vascular disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 2 | 0
Arthroscopy (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Open angle glaucoma (Eye disorders) | 1 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 50 mg (N=812) | Mirabegron 100 mg (N=820) | Tolterodine ER 4 mg (N=812)
Hypertension (Vascular disorders) | 74 | 80 | 78
Urinary tract infection (Infections and infestations) | 48 | 45 | 52
Dry mouth (Gastrointestinal disorders) | 23 | 19 | 70

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.